CLINICAL TRIAL: NCT05708950
Title: A Phase 1/2 Open-label Trial of KVA12123 Alone and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: A Clinical Trial of KVA12123 Treatment Alone and in Combination With Pembrolizumab In Advanced Solid Tumors (VISTA-101)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kineta Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VISTA-101; KEYNOTE-E67 (Other: Merck, Sharp & Dohme, LLC)
Record Dates: First submitted 2022-12-09; First posted 2023-02-01 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Solid Tumor; Melanoma; Carcinoma; Sarcoma; Lung Cancer; Prostate Cancer; Breast Cancer; Colo-rectal Cancer; Uterine Cancer; Pancreatic Cancer; Gastric Cancer; Esophageal Cancer; Thyroid Cancer; Ovarian Cancer; Kidney Cancer; Head and Neck Cancer
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma; Sarcoma; Lung Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Colonic Neoplasms; Uterine Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Thyroid Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KVA12123 Monotherapy Dose Escalation (Experimental): Part A will consist of dose escalation with KVA12123 administered as a single agent in participants with advanced solid tumors.
  Interventions: Drug: KVA12123 - Dose Escalation
- KVA12123 Plus Pembrolizumab Dose Escalation (Experimental): Part B will consist of dose escalation with KVA12123 administered in combination with a fixed dose of pembrolizumab.
  Interventions: Drug: KVA12123 Plus Pembrolizumab - Dose Escalation
- KVA12123 Monotherapy Dose Expansion (Experimental): Part C will consist of dose expansion with KVA12123 administered as a single agent at the RP2D in participants with advanced solid tumors.
  Interventions: Drug: KVA12123 - Dose Expansion
- KVA12123 Plus Pembrolizumab Dose Expansion (Experimental): Part D will consist of dose expansion with KVA12123 administered at the RP2D in combination with a fixed dose of pembrolizumab.
  Interventions: Drug: KVA12123 Plus Pembrolizumab - Dose Expansion

INTERVENTIONS:
Drug: KVA12123 - Dose Escalation — Ascending KVA12123 doses given as monotherapy by intravenous administration every 2 weeks of each 6-week cycle.
  Arms: KVA12123 Monotherapy Dose Escalation
Drug: KVA12123 Plus Pembrolizumab - Dose Escalation — Ascending KVA12123 doses given by intravenous administration every 2 weeks of each 6-week cycle in combination with a fixed dose of pembrolizumab administered once every 6 week cycle.
  Other Names: Keytruda
  Arms: KVA12123 Plus Pembrolizumab Dose Escalation
Drug: KVA12123 - Dose Expansion — KVA12123 administered at the RP2D by intravenous administration every 2 weeks of each 6 week cycle.
  Arms: KVA12123 Monotherapy Dose Expansion
Drug: KVA12123 Plus Pembrolizumab - Dose Expansion — KVA12123 administered at the RP2D by intravenous administration every 2 weeks in combination with a fixed dose of pembrolizumab administered once every 6 week cycle.
  Other Names: Keytruda
  Arms: KVA12123 Plus Pembrolizumab Dose Expansion

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of KVA12123 alone or combined with pembrolizumab in patients with advanced solid tumors. The main questions this study aims to answer are:

1. What is the safety of KVA12123 when administered alone and in combination with pembrolizumab to advanced cancer patients?
2. What is an appropriate dose of KVA12123 to administer alone and in combination with pembrolizumab to advanced cancer patients in future clinical trials?

Participants in this trial will be asked to:

1. Visit the clinical site every 1 - 2 weeks.
2. Receive KVA12123 every 2 weeks alone or in combination with pembrolizumab every 6 weeks.
3. Provide blood samples to evaluate drug levels in blood, drug safety and to explore the effects of each drug on the immune system.
4. Undergo scans every 6 weeks to test the effect of treatment on cancer progression.
5. Undergo other study procedures to evaluate drug safety and participant safety including physical exams, heart function tests, etc.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1/2, open-label, multicenter, dose escalation, and dose expansion study designed to evaluate the safety, tolerability, PK, immunogenicity, and tumor response of the investigational drug KVA12123 alone and in combination with pembrolizumab in adults with relapsed or refractory advanced solid tumors. The study will be conducted in 4 parts: Parts A and B will focus on dose escalation (single-agent and in combination), and Parts C and D will focus on dose expansion (single-agent and in combination).

Parts A (single-agent KVA12123) and B (KVA12123 + pembrolizumab) will comprise up to 10 dose escalation cohorts (6 for Part A and 4 for Part B) and treat 1-6 participants in each cohort to characterize the safety, tolerability, pharmacodynamics (PD), pharmacokinetics (PK) and preliminary tumor responses of study interventions. The objective of Parts A and B will be to determine a recommended Phase 2 dose (RP2D) for Parts C and D.

Parts C (single-agent KVA12123) and D (KVA12123 + pembrolizumab) will comprise up to 7 disease-specific dose expansion cohorts (2 for Part C and 5 for Part D), which will commence at the RP2D to further characterize the safety, tolerability, PD, PK, and preliminary tumor response of KVA12123 alone and in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to provide informed consent.
2. Be at least 18 years of age at the time of consent.
3. Has histologically or cytologically confirmed, locally advanced or metastatic solid tumor that has progressed or was non-responsive to standard of care therapy and for which no available curative therapy exists.
4. Has expected survival ≥16 weeks.
5. Presence of measurable disease by iRECIST.
6. Has an ECOG performance status score of 0 or 1.
7. Has adequate organ function within 10 days prior to the start of study treatment.
8. Has normal thyroid function or hypothyroid with stable supplementation.
9. Has consented to the collection of archival tissue prior to study treatment initiation.
10. Participants with prior exposure to systemic anticancer therapy including investigational agents following a 4-week washout period are eligible. Participants with prior small molecule targeted therapy or other short half-life drugs are eligible following a 2-week washout period.
11. Participants having prior curative radiation therapy completed 2 weeks prior to study drug administration or prior palliative radiation therapy to non-CNS disease completed at least 1 week prior to study drug administration are eligible.
12. HIV-infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease.
13. Participants with a history of HBV infection having durable HBsAg loss and undetectable serum HBV DNA no longer requiring treatment are eligible.
14. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening and participants have completed curative antiviral therapy.
15. Post-menopausal women and surgically sterile men and women are permitted.
16. Patients of childbearing potential are permitted to participate under the following conditions:

    1. Must have negative urine pregnancy test result within 72 hrs prior to the first dose of any study drug
    2. Must agree not to become pregnant during the study and for 120 days after the final dose of any study drug
    3. Must agree not to breastfeed or donate ova, starting at time of informed consent and continuing through 120 days after the final dose of any study drug
    4. If sexually active in a way that could lead to pregnancy, must consistently use 2 acceptable methods of birth control (contraception), at least 1 of which must be highly effective starting at time of informed consent and continuing throughout the study and for 120 days after the final dose of any study drug.
17. Patients who can father children are permitted to participate under the following conditions:

    1. Must agree not to donate sperm starting at the time of informed consent and continuing throughout the study period and for 120 days after the final dose of any study drug
    2. If sexually active with a person of childbearing potential in a way that could lead to pregnancy, must consistently use 2 acceptable methods of birth control (contraception), at least 1 of which must be highly effective starting at the time of informed consent and continuing throughout the study and for 120 days after the final dose of any study drug
    3. If sexually active with a person who is pregnant or breastfeeding, must consistently use a condom starting at time of informed consent and continuing throughout the study and for 120 days after the final dose of any study drug.
18. Must be willing and able to comply with the trial procedures and the follow-up schedule.

Exclusion Criteria

1. Untreated CNS metastatic disease, leptomeningeal disease, or cord compression.
2. Concurrent cancer other than disease under study requiring systemic treatment. Participants with basal cell or squamous cell skin cancer treated with curative intent, carcinoma in-situ of the cervix or breast treated with curative intent, RAI stage 0 Chronic Lymphocytic Leukemia, monoclonal gammopathy of undetermined significance, superficial bladder cancer or very low and low risk prostate cancer (localized Gleason score ≤ 6) under active surveillance are eligible.
3. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
4. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg QD of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
5. History of (non-infectious) pneumonitis/interstitial lung disease (ILD) that required steroids or current pneumonitis/ILD.
6. Prior treatment with VISTA-targeted therapy.
7. Prior history of allogeneic, solid organ or stem cell transplant, or adoptive T-cell transplant.
8. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, LAG-3, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related adverse event (irAE).
9. Active known or suspected autoimmune disease that has required systemic treatment within the past year. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Prior systemic anticancer therapy, including investigational agents, within 4 weeks of treatment. Participants with prior small molecule targeted therapy or other short half-life drugs are eligible following a 2-week washout period.
11. Has received prior radiation therapy within 2 weeks of start of study treatment or has a history of radiation pneumonitis.
12. Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study treatment.
13. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
14. Any requirement for daily supplemental oxygen.
15. Any condition requiring systemic treatment with corticosteroids (>10 mg QD prednisone equivalents) or other immunosuppressive medications within 14 days before the first dose of study drug.
16. Serious or poorly controlled cardiovascular disease.
17. Chronic hepatitis B or C.
18. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
19. Has an active infection requiring systemic therapy.
20. Known active or latent tuberculosis.
21. If the participant had major surgery, must have recovered adequately from the procedure and/or any complications.
22. Toxicities arising from prior cancer therapy that have not resolved to Grade 1 or baseline.
23. Red blood cell or platelet infusion within the preceding 2 weeks.
24. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
25. Known hypersensitivity to any excipient contained in the drug formulation of KVA12123.
26. Any significant history of drug allergy as assessed by the investigator.
27. Positive urine pregnancy test within 72 hrs of study drug administration.
28. Participants who are breastfeeding, pregnant, or planning to become pregnant from time of informed consent until at least 120 days after final dose of study drug.
29. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study.
30. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
31. Inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through study completion, an average of 1 year
  Type and frequency of adverse events as assessed by CTCAE v4.0.
AEs related to study drug | Through study completion, an average of 1 year
  Type and frequency of treatment related adverse events as assessed by CTCAE v4.0.
Recommended Phase 2 dose (RP2D) or maximum tolerated dose (MTD) | Through study completion, an average of 1 year
  Recommended Phase 2 dose (RP2D) or maximum tolerated dose (MTD) of KVA12123 when administered alone and in combination with pembrolizumab in participants with advanced solid tumors (milligrams or milligrams/kilogram).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of KVA12123 (Cmax) | Through study completion, an average of 1 year
  maximum serum concentration (micrograms/milliliter [mL])
Pharmacokinetic (PK) profile of KVA12123 (Cmin) | Through study completion, an average of 1 year
  trough serum concentration (micrograms/mL)
Pharmacokinetic (PK) profile of KVA12123 (tmax) | Through study completion, an average of 1 year
  time to maximum serum concentration (hours)
Pharmacokinetic (PK) profile of KVA12123 (AUC) | Through study completion, an average of 1 year
  Area under the concentration-time curve (microgram*mL/hour)
Pharmacokinetic (PK) profile of KVA12123 (t1/2) | Through study completion, an average of 1 year
  Elimination half life (hours)
Pharmacokinetic (PK) profile of KVA12123 (Vd) | Through study completion, an average of 1 year
  Volume of distribution (milliliter or liter)
Pharmacokinetic (PK) profile of KVA12123 (Cl) | Through study completion, an average of 1 year
  Clearance (mL/hour)
Concentration of anti-KVA12123 antibodies in serum | Through study completion, an average of 1 year
  Change from baseline in anti-KVA12123 antibodies in serum (antibody concentration per mL)
Number of participants with progressive disease following treatment with KVA12123 | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with progressive disease following treatment with KVA12123 in combination with pembrolizumab | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with stable disease following treatment with KVA12123 | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with stable disease following treatment with KVA12123 plus pembrolizumab | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with partial response following treatment with KVA12123 | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with partial response following treatment with KVA12123 plus pembrolizumab | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with complete response following treatment with KVA12123 | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.
Number of participants with complete response following treatment with KVA12123 plus pembrolizumab | Through study completion, an average of 1 year
  Investigator assessment of radiographic imaging according to iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Guillaudeux, PhD, Study Director — Kineta Inc.
Locations (6):
- United States (6):
  - UCLA Health (Santa Monica Cancer Care), Santa Monica, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Sarasota, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No